CLINICAL TRIAL: NCT05652946
Title: Clinicians, Academics, Industry, and Insurance Collaborate to Assess Cost-Effectiveness and Functional Outcomes Using Advanced Rehabilitation Technology
Brief Title: IISART (International Industry Society of Advanced Rehabilitation Technology) Advanced Rehabilitation Technology Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rehabilitation Hospital of Overland Park (Industry)
Collaborators: Discovery Statistics (Unknown)
Responsible Party: Principal Investigator, Brett Schoen, Medical Director, Rehabilitation Hospital of Overland Park
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PH750
Record Dates: First submitted 2022-11-14; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Neurologic Disorder
Keywords: Advanced Rehabilitation Technology; Therapeutic Device; Robotic Rehabilitation Research; Health Economics; Functional Outcomes
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: One group receives inpatient rehabilitation with advanced rehabilitation technology and one group receives inpatient traditional rehabilitation without advanced rehabilitation technology.
Who Masked: Outcomes Assessor
Masking Description: Masked/blinded outpatient therapists will perform outcome assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Inpatient Rehabilitation with ART (Experimental): Inpatient rehabilitation with advanced rehabilitation technology
  Interventions: Device: Tyromotion, Fourier Intelligence, Thera-Trainer, EKSO Bionics
- Inpatient Rehabilitation without ART (Active Comparator): Inpatient rehabilitation without advanced rehabilitation technology
  Interventions: Other: Standard inpatient rehabilitation therapy

INTERVENTIONS:
Device: Tyromotion, Fourier Intelligence, Thera-Trainer, EKSO Bionics — Participants to receive at least 5 sessions with advanced rehabilitation technology including at least one, or multiple, of the following devices: Amadeo, Diego, Myro, Arm Motus EMU, Pelma Motus, Tigo, Balo, EKSO NR. Sessions are 45 (+/- 5) minutes
  Arms: Inpatient Rehabilitation with ART
Other: Standard inpatient rehabilitation therapy — Standard inpatient rehabilitation therapy without advanced rehabilitation technology
  Arms: Inpatient Rehabilitation without ART

SUMMARY:
A pre-post, randomized control trial comparing cost-effective and functional outcomes of participants with neurological diagnoses using robotic devices and advanced technology during inpatient rehabilitation to the outcomes of control participants without the use of robotic devices and advanced technology during rehabilitation. We aim to show at least similar inpatient rehabilitation outcomes and improved health economics in participants with neurological diagnoses by using robotic devices and advanced technology to increase the intensity and dose of rehabilitation.

DETAILED DESCRIPTION:
Many previous trials have shown equivalency of outcomes when comparing use of a robotic device vs standard therapy. Most often, the intensity was held equal between the two groups. However, robotic devices can greatly improve the intensity and dose of upper and lower extremity rehabilitation, while reducing therapist burden. Moreover, the outcome measures used in these previous studies were not specific to the task practiced in the device, or the task was not practiced outside of the device. This study provides robotic devices and advanced technology as part of the overall therapy plan and will include outcome measures based on individual participant return to community, in addition to health economic and functional measures. The rationale to use multiple robotic devices and advanced technology as part of rehabilitation is to improve quality of life/return to community as well as health economics and therapy outcomes.

Hypotheses:

1. Assuming no difference in functional outcomes across groups, participants with neurological diagnoses receiving inpatient rehabilitation with robotic devices and advanced technology will show better quality of life/return to community and health economics outcomes (superiority hypothesis) compared to controls who do not receive rehabilitation with robotic devices or similar advanced technology.
2. Participants with neurological diagnoses receiving inpatient rehabilitation with robotic devices and advanced technology will show functional outcomes at least as good as (non-inferiority hypothesis) those compared to controls who do not receive rehabilitation with robotic devices or similar advanced technology

ELIGIBILITY:
Inclusion Criteria:

1. Currently admitted for inpatient rehabilitation at Rehabilitation Hospital Overland Park with neurological diagnosis.
2. At least 18 years of age.
3. Predicted length of stay to be at least 7 days.
4. Able to tolerate upright sitting without orthostatic hypotension for upper extremity, cycling, and sitting balance devices AND/OR able to tolerate upright standing for at least 15 minutes without orthostatic hypotension for walking and standing balance devices.
5. Able to fit into at least one device.
6. Screened and cleared by a physician.
7. Cognitively intact to communicate pain and/or need to stop session, and able to follow simple commands.

Exclusion Criteria:

1. Current or history of other medical conditions that could affect the outcome measures.
2. Currently involved in another intervention study.
3. Any absolute contraindication listed for each device used.
4. Any pre-existing physical or medical condition that the Physiatrist determines would significantly limit a patient's ability to benefit from or continue in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-10-17 (Estimated); Study Completion 2025-01-17 (Estimated)

PRIMARY OUTCOMES:
Neuro-QOL | Through study completion, an average of 2 years
  Neuro-QOL battery: Ability to Participate in Social Roles and Activities, Satisfaction with Social Roles and Activities, Positive Affect and Well-Being

SECONDARY OUTCOMES:
Length of stay/# of visits | Through study completion, an average of 2 years
  Length of stay/# of visits
Total cost of care (TCOC) | Through study completion, an average of 2 years
  Total cost of care (TCOC)
Cost of caregiver burden | Through study completion, an average of 2 years
  Cost of caregiver burden
Discharge disposition | Through study completion, an average of 2 years
  Discharge disposition
Return to work/school/volunteer | Through study completion, an average of 2 years
  Return to work/school/volunteer
Return to Recreation | Through study completion, an average of 2 years
  Return to Recreation
Areas of pain | Through study completion, an average of 2 years
  Visual analog scale for patient report of pain
Spasticity | Through study completion, an average of 2 years
  Visual analog scale for patient report of spasticity
Section GG scores | Through study completion, an average of 2 years
  Functional Abilities and Goals
10 Meter Walk Test | Through study completion, an average of 2 years
  Gait speed
Functional Ambulation Category | Through study completion, an average of 2 years
  Walking ability
Functional Reach | Through study completion, an average of 2 years
  Functional balance
Tinetti-Fall Efficacy Scale | Through study completion, an average of 2 years
  Patient confidence regarding falls
Manual muscle test (MMT) | Through study completion, an average of 2 years
  To test strength of upper and lower extremities
Range of Motion (ROM) | Through study completion, an average of 2 years
  To test range of motion of upper and lower extremity joints
Quick DASH (Disabilities of the Arm, Shoulder, and Hand) | Through study completion, an average of 2 years
  Upper extremity function

OTHER OUTCOMES:
Goal attainment scale (GAS) | Through study completion, an average of 2 years
  Patient report of goal setting

CONTACTS AND LOCATIONS:
Overall Officials: Brett Schoen, MD, Principal Investigator — Rehabilitation Hospital of Overland Park
Locations (1):
- Rehabilitation Hospital of Overland Park, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spiess MR, Steenbrink F, Esquenazi A. Getting the Best Out of Advanced Rehabilitation Technology for the Lower Limbs: Minding Motor Learning Principles. PM R. 2018 Sep;10(9 Suppl 2):S165-S173. doi: 10.1016/j.pmrj.2018.06.007. PMID 30269803